CLINICAL TRIAL: NCT00631254
Title: Modulation of the CysLT1-r Expression Following Allergen Exposure in Non Asthmatic Subjects With Allergic Rhinitis and Mild Allergic Asthmatic Subjects Using the Induced Sputum Technique.
Brief Title: CysLT1-r Expression Following Allergen Exposure in Asthma and Allergic Rhinitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Louis-Philippe Boulet, Laval Hospital
Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P1179
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2008-05-12 (Estimated); Status verified 2007-11

CONDITIONS: Asthma; Allergic Rhinitis
MeSH Terms: conditions — Asthma; Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Conventional allergen challenge: increasing allergen doses given by nebulisation through the mouth and stopped when a 20% fall in forced expiratory volume in one second is obtained.
  Low dose allergen challenge: very low allergen doses given by nebulisation through the mouth. No more than a 5% fall in forced expiratory volume in one second.
  Nasal allergen challenge: One drop of increasing allergen doses on nasal mucosa.
  Interventions: Procedure: Allergen challenge
- 2 (Active Comparator): Low dose allergen challenge: very low allergen doses given by nebulisation through the mouth. No more than a 5% fall in forced expiratory volume in one second.
  Nasal allergen challenge: One drop of increasing allergen doses on nasal mucosa.
  Interventions: Procedure: Allergen challenge

INTERVENTIONS:
Procedure: Allergen challenge — Conventional allergen challenge: increasing allergen doses given by nebulisation through the mouth and stopped when a 20% fall in forced expiratory volume in one second is obtained.
  Low dose allergen challenge: very low allergen doses given by nebulisation through the mouth. No more than a 5% fall in forced expiratory volume in one second.
  Nasal allergen challenge: One drop of increasing allergen doses on nasal mucosa.
  Arms: 1
Procedure: Allergen challenge — Low dose allergen challenge: very low allergen doses given by nebulisation through the mouth. No more than a 5% fall in forced expiratory volume in one second.
  Nasal allergen challenge: One drop of increasing allergen doses on nasal mucosa.
  Arms: 2

SUMMARY:
Cysteinyl leukotrienes (CysLTs) play an important role in asthma. CysLTs exert most of their bronchoconstrictive and pro-inflammatory effects through activation of the CysLT1-r. As allergic rhinitis appears to be a predisposing factor in the development of asthma and as CysLT-receptors seem to be implicated in the first steps of asthma manifestations, we think it would be of interest to determine if the CysLT1-r is a key mediator in the progression from allergic rhinitis to asthma. We believe it would be interesting to study the expression of the CysLT1-r

Our goal is to assess baseline, as well as variations following allergen bronchoprovocations, in the expression of the CysLT1-r in mild asthmatic subjects compared with non asthmatic subjects with allergic rhinitis.

Our hypothesis is that there will be a higher baseline expression of the CysLT1-r in asthmatic subjects compared with allergic rhinitis subjects and that allergen bronchoprovocations will induce an increase in the expression of the CysLT1-r in both groups.

DETAILED DESCRIPTION:
We will recruit mild allergic asthmatic subjects and non asthmatic subjects with allergic rhinitis. On a baseline visit, allergy skin prick tests, spirometry, methacholine bronchoprovocation and induced sputum (IS) with differential leukocyte count will be obtained.

In a second step, mild asthmatic subjects will undergo conventional bronchial allergen challenge. IS will be obtained at 6h (corresponding to the late asthmatic response) and 24h following the challenge. The rhinitic subjects and asthmatic subjects will undergo a 4-day low dose allergen bronchial challenge as well as a nasal allergen challenge. Sputum samples will be obtained following days 2 and 4 of the low dose challenge and one week later, and 24h following nasal challenge.

Induced sputum will be analyzed for differential cell count. Total mRNA will be extracted from IS cells and used for RT-PCR.

ELIGIBILITY:
Inclusion Criteria:

* To have a positive reaction to one or more allergen on prick tests.
* Non smokers
* No respiratory track infection for at least one month prior to the study.
* Asthmatic subjects using only inhaled beta-2 agonists on an as needed basis for their asthma treatment.
* Asthmatic subjects with a history of asthma of at least 6 months.
* Asthmatic subjects with PC20 methacholine lower or equal to 8 mg/ml.
* Allergic rhinitic subjects never experienced any asthma symptoms or took any asthma medication in the past.
* Allergic rhinitic subjects with a PC20 methacholine higher than 16 mg/ml.

Exclusion Criteria:

* Smokers or ex smokers less than 6 months or more than 10 pack-years.
* Asthmatic subjects using or used in the past 3 months inhaled or oral corticosteroids.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-10; Primary Completion 2009-01 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Change in CysLT1-r following allergen challenge | At 7h and 24h following conventional challenge

SECONDARY OUTCOMES:
Change in CysLT1-r following low dose allergen challenge | At 2 and 4 days of challenge
Difference in CysLT1-r expression in asthma and allergic rhinitis | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — Hopital Laval
Locations (1):
- Centre de recherche de l'Hopital Laval, Québec, Quebec, Canada